CLINICAL TRIAL: NCT05556902
Title: Therapeutic Mechanisms of Epidural Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Marshall Holland, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300009200; UAB (Other: UAB)
Record Dates: First submitted 2022-09-02; First posted 2022-09-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Blood Pressure; Low Back Pain; Hypertension
Keywords: Spinal Cord Stimulation; Epidural Spinal Cord Stimulation; SCS; Arterial Blood Pressure
MeSH Terms: conditions — Low Back Pain; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Patients that proceed with permanent implantation of a spinal cord stimulator.
  Interventions: Device: Permanent Epidural Spinal Cord Stimulation
- Control (No Intervention): Patients who do not proceed with permanent implantation of a spinal cord stimulator.

INTERVENTIONS:
Device: Permanent Epidural Spinal Cord Stimulation — Permanent Spinal Cord Stimulation implanted in participants undergoing routine care for management of chronic neuropathic pain.
  Arms: Treatment

SUMMARY:
The purpose of this study in patients undergoing routine care epidural spinal cord stimulation (SCS) is to determine 1) whether SCS reduces arterial blood pressure (BP) in patients which chronic low back pain and hypertension, 2) whether higher baseline BP (i.e., hypertension) predicts reductions in pain following SCS, and finally 3) whether different SCS waveforms elicits stimulus-evoked compound action potentials (ECAPs) in spinal cord and at the cortex (electroencephalography, and magnetoenchphalography).

DETAILED DESCRIPTION:
The purpose of this study in patients undergoing routine care epidural spinal cord stimulation (SCS) is to determine 1) whether SCS reduces arterial blood pressure (BP) in patients which chronic low back pain and hypertension, 2) whether higher baseline BP (i.e., hypertension) predicts reductions in pain following SCS, and finally 3) whether different SCS waveforms elicits stimulus-evoked compound action potentials (ECAPs) in spinal cord and at the cortex (electroencephalography, and magnetoenchphalography).

The Investigators will identify patients with chronic pain who are scheduled for SCS implant at the University of Alabama at Birmingham for management of chronic neuropathic pain as part of routine care. The research team will assess BP with an arm cuff arm cuff before and after the implant among patients providing written informed consent.

The Investigators' central clinical hypothesis is that SCS decreases blood pressure in patients with chronic pain and comorbid hypertension. The Investigators further hypothesize that the SCS will improve serological markers of sympathetic nerve activity and kidney function, possibly due to reductions in spinal cord sympathetic nerve activity. A secondary hypothesis is that higher baseline blood pressure predicts larger reductions in blood pressure following SCS implant.

Additionally, this project seeks to expand knowledge on therapeutic mechanisms of SCS via recording electrophysiological responses at the spinal cord (via adjacent, unused SCS contacts) and from EEG scalp recordings over the cerebral cortex.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, age 18-89
2. Chronic pain for more than 3 months
3. Willing to visit a research lab
4. Willing to undergo a blood draw
5. Able to provide written informed consent

Exclusion Criteria

1. History of neurological disease (e.g., dementias, Parkinson's)
2. History of stroke
3. Current diagnosis of cancer
4. Subject is unwilling or unable to comply with the protocol

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Pressure Change | Baseline (1 week pre-op)
  The research team will assess systolic and diastolic blood pressure with an arm cuff.
Arterial Blood Pressure Change | Visit 2 (4-6 weeks post-op)
  The research team will assess systolic and diastolic blood pressure with an arm cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Holland, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT05556902/SAP_000.pdf